CLINICAL TRIAL: NCT06091787
Title: Effect of Ursodeoxycholic Acid Supplementation on Liver Regeneration on Right Lobe Donor Hepatectomy: An Open Label Randomised Trial
Brief Title: Effect of Ursodeoxycholic Acid Supplementation on Liver Regeneration on Right Lobe Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2023/104/MA01
Record Dates: First submitted 2023-10-05; First posted 2023-10-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Liver Regeneration; Ursodeoxycholic Acid; Partial Liver Resection
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Open label randomised controlled trial with 2 groups. One group receiving Tablet Ursodeoxycholic acid and the other group not receiving standard medical therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm (Experimental): This group will recieve Tab Ursodeoxycholic acid 450mg twice daily from the day after donor hepatectomy till post operative day 10.
  Interventions: Drug: Ursodeoxycholic acid
- Control Arm (Active Comparator): This group will receive standard medical therapy following donor hepatectomy.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Ursodeoxycholic acid — Tablet Ursodeoxycholic acid 450mg per orally twice daily from Post operative day 1 to post operative day 10.
  Arms: Study Arm
Other: Standard Medical Treatment — Standard Medical Treatment
  Arms: Control Arm

SUMMARY:
The goal of this open label randomized trial is to understand the role of oral ursodeoxycholic acid(UDCA) supplementation in the liver regeneration (in terms of liver function and anatomical growth) following right lobe donor hepatectomy. The main question it aims to answer are:

* Does Ursodeoxycholic acid supplementation on patients undergoing donor hepatectomy improve anatomical liver regeneration after partial hepatectomy as compared to control group.
* Does ursodeoxycholic acid improve liver regeneration in terms of liver function tests and biomarkers of liver regeneration(HGF, IL6, TNF Alpha, AFP, TGF Beta) as compared to control group.

DETAILED DESCRIPTION:
This open label randomized control study aims to analyze the effect of ursodeoxycholic acid supplementation on liver regeneration following a right donor hepatectomy. All eligible live donors who undergo right donor hepatectomy during the study period will be included in the study and randomized into two groups. One group will receive Tab. UDCA 450mg twice daily for 10 days and the other group will not receive Tab UDCA. Live donors who are not willing to participate in the study, have hypersensitivity to UDCA or have used Tab UDCA in the past 2 weeks, will be excluded from the study. All live donors will be screened in the pre-operative period in the outpatient department.

Pre- operative, intra-operative and post-operative data will be collected from medical records, electronic hospital information system (HIS) and radiological images collected from the hospital Picture archiving and communication system(PACS). The enrolled subjects will be followed up till for a period of 14 days after the donor hepatectomy till Non contrast CT Abdomen is done and regenerated liver volumes are analyzed. The anatomic(volumetric), functional(liver function tests) and regenerative biomarkers( HGF, TNF-Alpha, IL6, AFP, TGF-Beta) will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All live donors undergoing Right Donor Hepatectomy in ILBS from ethical board clearance to December 2024 in the Department of HPB Surgery and Liver Transplantation, Institute of Liver and Biliary Sciences, New Delhi

Exclusion Criteria:

* Negative consent
* Hypersensitivity to UDCA
* Past history of UDCA use in the last two weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Regenerated liver volume on Post-operative Day 14 between two groups. | 14 days after operation
  * This will be measured by a non contrast CT Abdomen and the size of the regenerated liver after hepatectomy will be measured in millilitres
  * This value will be measured in both groups to identify a difference in the intervention group (getting UDCA) versus the control group ( standard medical therapy)
Regenerated liver volume on Post-operative Day 7 between two groups. | 7 days after operation
  * This will be measured by a non contrast CT Abdomen and the size of the regenerated liver after hepatectomy will be measured in millilitres
  * This value will be measured in both groups to identify a difference in the intervention group (getting UDCA) versus the control group ( standard medical therapy)
Percentage of Total Liver Volume Restored on Post-operative Day 7 between two groups. | 7 days after operation
  The percentage of Total liver volume restored on Post operative day 7 compared to the pre-operative total liver volume, between two groups.
Percentage of Liver Volume restored on Post-operative Day 14 between two groups. | 14 days after the operation
  Percentage of liver volume restored on on Post operative day 14, compared to pre-operative total liver volume, between two groups.
Absolute Liver Volume growth on Day 7 | 7 days after the operation
  Pre-operative remnant liver volume subtracted from regenerated liver volume on Post-operative day 7, between both groups.
Absolute Liver volume growth on day 14 | 14 days after the operation
  Pre-operative remnant liver volume subtracted from regenerated liver volume on Post-operative day 14, between both groups.
Regeneration Velocity on Post operative day 14, between both groups | 14 days after the operation
  Rate of regeneration of liver(g/day), denoted by subtracting pre-operative remnant liver volume from regenerated liver volume on post operative day 14, divided by 14.

SECONDARY OUTCOMES:
Total bilirubin | Post-operative day 1-7, 10 and 14
  serum total bilirubin versus control group
Direct bilirubin | Post-operative day 1-7, 10 and 14
  serum Direct bilirubin versus control group
Alanine Aminotransferase(ALT) | Post-operative day 1-7, 10 and 14
  serum ALT versus control group
Aspartate Aminotransferase(AST) | Post-operative day 1-7, 10 and 14
  serum AST versus control group
Serum Alkaline Phosphatase(SAP) | Post-operative day 1-7, 10 and 14
  serum SAP versus control group
Serum Gamma Glutamyl Transferase(GGT) | Post-operative day 1-7, 10 and 14
  serum SAP versus control group
Serum Albumin | Post-operative day 1-7, 10 and 14
  serum Albumin versus control group
International normalized ratio(INR) | Post-operative day 1-7, 10 and 14
  INR versus control group
Post hepatectomy liver failure(PHLF) | Post operative day 1-14
  Grade of PHLF as per ISGLS criteria and 50/50 criteria
Abdominal Drain removal | Post operative day 1-14
  Day of abdominal drain removal
Post-operative ascites | Post operative day 1-14
  Volume of ascites
Post-operative complications | Post operative day 1-14
  Grade of post-operative complications as per Clavien-Dindo classification
Markers of liver regeneration - Serum TNF Alpha | Pre-op Baseline, Post-operative Day 1, Post-operative Day 3, Post-operative Day7
  Serum TNF Alpha vs in Control group
Markers of liver regeneration - Serum IL6 | Pre-op Baseline, Post-operative Day 1, Post-operative Day 3, Post-operative Day 7
  Serum IL6 vs in Control group
Markers of liver regeneration - Serum Alpha Fetoprotein | Pre-op Baseline, Post-operative Day 1, Post-operative Day 3, Post-operative Day 7
  Serum Alpha Fetoprotein vs in Control group
Markers of liver regeneration - TGF Beta | Pre-op Baseline, Post-operative Day 1, Post-operative Day 3, Post-operative Day 7
  TGF Beta vs in Control group
Markers of liver regeneration - Hepatocyte growth factor in blood | Pre-op Baseline , Post-operative Day 1, Post-operative Day 3, Post-operative Day 7
  Hepatocyte growth factor vs in Control group

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Rn Mohapatra, MBBS,MS, MCh, Study Chair — Institute of Liver and Biliary Sciences, New Delhi
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No